CLINICAL TRIAL: NCT00172224
Title: Dynamic MR Study in Evaluating the Vertebral Bone Marrow Perfusion and Its Related Research
Brief Title: Dynamic Magnetic Resonance (MR) Study in Evaluating the Vertebral Bone Marrow Perfusion and Its Related Research
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 32244; NSC 91-2314-B-002-395; NSC 92-2314-B-002-172
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Osteoporosis; Fractures, Compression
Keywords: osteoporosis; compression fracture; bone marrow perfusion; MR spectroscopy; hormone therapy
MeSH Terms: conditions — Osteoporosis; Fractures, Compression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- osteoporosis

SUMMARY:
The etiology and pathogenesis of osteoporosis has been extensively discussed. The relationship between bone blood circulation and the formation of bony trabeculae has been less understood. There is plenty of indirect evidence highly suggestive of the correlation between these two factors, such as: the number of blood vessels in the per unit area of the bone marrow was decreased in the osteoporotic bone, indicating the possible role of a microvascular defect in the pathogenesis of osteoporosis.

Furthermore, the bone mineral density in severe arteriosclerotic patients was lower than in the less affected subjects. In a large scale epidemiologic study, diminished bone mineral density was strongly associated with increased deaths from stroke. Osteopenia was also associated with an increased risk of stroke. These reports highly suggest the effect of ischemia on bone metabolism and make the investigators more interested in further investigation.

A dynamic contrast-enhanced magnetic resonance (MR) study was used recently in evaluating the blood perfusion of bone tumors. This method also has a strong correlation with the microsphere blood flow measurements. The investigator (T.F. Shih) used the dynamic MR in her recent two researches:

1. To differentiate benign versus malignant spinal compression fractures.
2. To evaluate the blood perfusion of non-fractured, normal-appearing vertebral bodies and find its significant correlation with aging and sex.

The alterations of bone marrow perfusion are synchronous with the changes of bone mineral density. Thus, based on the investigators' previous research work, they propose to further explore the relationship between bone marrow perfusion and bone mineral density in different age groups.

DETAILED DESCRIPTION:
The etiology and pathogenesis of osteoporosis has been extensively discussed. The relationship between bone blood circulation and the formation of bony trabeculae has been less understood. There is plenty of indirect evidence highly suggestive of the correlation between these two factors, such as: the number of blood vessels in the per unit area of the bone marrow was decreased in the osteoporotic bone, indicating the possible role of a microvascular defect in the pathogenesis of osteoporosis.

Furthermore, the bone mineral density in severe arteriosclerotic patients was lower than in the less affected subjects. In a large scale epidemiologic study, diminished bone mineral density was strongly associated with increased deaths from stroke. Osteopenia was also associated with an increased risk of stroke. These reports highly suggest the effect of ischemia on bone metabolism and make the investigators more interested in further investigation.

A dynamic contrast-enhanced magnetic resonance (MR) study was used recently in evaluating the blood perfusion of bone tumors. This method also has a strong correlation with the microsphere blood flow measurements. The investigator (T.F. Shih) used the dynamic MR in her recent two researches:

1. To differentiate benign versus malignant spinal compression fractures.
2. To evaluate the blood perfusion of non-fractured, normal-appearing vertebral bodies and find its significant correlation with aging and sex.

The alterations of bone marrow perfusion are synchronous with the changes of bone mineral density. Thus, based on the investigators' previous research work, they propose to further explore the relationship between bone marrow perfusion and bone mineral density in different age groups.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects
* Elder subjects with osteoporosis

Exclusion Criteria:

* History of malignancy or infection

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects with osteoporosis
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Ting-Fang Shih, M.D., Principal Investigator — Department of Medical Image, National Taiwan University Hospital
Locations (1):
- Tiffany Ting-Fang Shih, Taipei, Taiwan